CLINICAL TRIAL: NCT06748105
Title: Dapagliflozin as Prophylaxis for Glucocorticoid-Induced Hyperglycemia: Phase II Randomized Clinical Trial
Brief Title: Dapagliflozin as Prophylaxis for Glucocorticoid-Induced Hyperglycemia
Acronym: DAPACOID
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lauro Fabián Amador Medina (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor-Investigator, Lauro Fabián Amador Medina, Principal Investigator, Coordinación de Investigación en Salud, Mexico
Organization: Coordinación de Investigación en Salud, Mexico (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R-2024-1001-047
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Dapagliflozin (Forxiga); Hyperglycaemia; Glucocorticoid
Keywords: dapagliflozin; hyperglycaemia; glucocorticoid
MeSH Terms: conditions — Hyperglycemia | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Protocol Design:
  Participants will be randomized 1:1, with group assignments known to all. Dapagliflozin (10 mg/day) will be administered orally within 12 hours of glucocorticoid dosing. Adherence will be ensured through patient/family training and nursing reports.
  Intervention Monitoring:
  Daily glucose levels will be assessed via preprandial capillary measurements (three shifts) and fasting central glucose (6-8 hours fasting). Standard glycemic monitoring (SGM) will also be performed.
  Definitions for Objectives:
  Hyperglycemia (HIG): ≥2 readings ≥140 mg/dL (7.8 mmol/L) in 24 hours. Hyperglycemic Crisis (HC): ≥2 readings ≥180 mg/dL (>10 mmol/L) in 24 hours. If insulin or other antidiabetic treatments are initiated, they will be allowed alongside dapagliflozin in the intervention arm, with their use documented.
  Safety Monitoring:
  Adverse events will be recorded for all groups. Follow-up will continue until discharge, 10 days, or whichever occurs first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Participants in this arm will receive dapagliflozin (10 mg/day) administered orally. The dose will be synchronized with glucocorticoid administration, with a maximum allowable time difference of 12 hours. Patients and their families will be trained in self-administration, and adherence will be monitored through nursing service reports.
  Interventions: Drug: Dapagliflozin (DAPA)
- Standard Monitoring Arm (Active Comparator): Participants will undergo standard glycemic monitoring (SGM), including preprandial capillary glucose measurements during three daily shifts and fasting central glucose assessments (6-8 hours fasting).
  Interventions: Drug: Dapagliflozin (DAPA)

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Participants will receive 10mg/day of dapagliflozin orally. The administration will occur within a "synchronous" range, meaning that the time difference between dapagliflozin administration and glucocorticoid administration should not exceed 12 hours.

SUMMARY:
The goal of this clinical trial is to investigate whether dapagliflozin can help prevent glucocorticoid-induced hyperglycemia (GIH) in hospitalized patients requiring high-dose glucocorticoids (GCs). This trial will also assess the safety of dapagliflozin when used alongside GCs. The main questions the trial aims to answer are:

Does dapagliflozin reduce the incidence of GIH in patients receiving high-dose GCs? What side effects or adverse events occur in patients taking dapagliflozin alongside high-dose GCs? Researchers will compare dapagliflozin to standard glucose monitoring (SGM) to determine if dapagliflozin is effective in preventing GIH in patients receiving high doses of GCs.

Participants will:

Take dapagliflozin (10 mg/day) or undergo standard glucose monitoring during their hospital stay.

Visit the hospital for regular check-ups and glucose testing during their treatment.

Record their glucose levels multiple times a day and report any adverse events they experience.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the efficacy and safety of dapagliflozin in preventing glucocorticoid-induced hyperglycemia (GIH) in hospitalized patients who require high-dose glucocorticoid (GC) treatment. GCs are commonly used in clinical practice for their potent anti-inflammatory and immunosuppressive properties, but they are also a major cause of medication-induced hyperglycemia, particularly when administered at high doses.

The hypothesis of this trial is that dapagliflozin, a sodium-glucose cotransporter-2 (SGLT2) inhibitor, may reduce the incidence of GIH by counteracting the metabolic disturbances caused by GCs. Dapagliflozin works by inhibiting the SGLT2 protein, which is responsible for glucose reabsorption in the kidneys. By inhibiting this protein, dapagliflozin promotes glucose excretion in the urine, helping to reduce blood glucose levels. This mechanism is particularly relevant in the context of GIH, as GCs can impair insulin secretion, promote hepatic gluconeogenesis, and increase peripheral insulin resistance.

The primary aim of the study is to compare the incidence of GIH in patients receiving dapagliflozin versus those undergoing standard glucose monitoring (SGM) while on high-dose GCs. Secondary objectives include assessing the cumulative incidence of GIH days, the number of hyperglycemic crises, and the need for insulin therapy. The study also evaluates the safety profile of dapagliflozin, particularly focusing on any adverse events associated with its use in this population. The adverse effects of high-dose GCs will also be reported to provide a broader context for understanding the potential risks of treatment.

This randomized, open-label, controlled clinical trial will enroll hospitalized patients aged 18 and older who require high-dose GC therapy (prednisone equivalents >30 mg/day). The study will be conducted at the High Specialty Medical Unit, Hospital of Specialties No. 1, National Medical Center of Bajío, Mexican Institute of Social Security. Participants will be randomly assigned to one of two groups: the dapagliflozin group (10 mg/day) or the control group receiving standard glucose monitoring (SGM).

Both groups will undergo routine glucose monitoring through capillary glucose checks (three times daily) and fasting central glucose assessments. The study will be conducted during the patients' hospitalization, and participants will be followed until discharge or up to 10 days, whichever occurs first. The dosing schedule for dapagliflozin will ensure it is administered synchronously with the GC dose (within 12 hours of GC administration).

Additionally, data regarding the incidence of insulin therapy use, as well as the incidence and duration of hyperglycemic crises (defined as ≥2 persistent glucose readings ≥180 mg/dL within 24 hours), will be carefully recorded and analyzed. Adverse events will be monitored throughout the study, with particular attention to renal function, as SGLT2 inhibitors have been associated with potential renal side effects in some patient populations.

The statistical analysis will be based on comparing the two treatment arms for the incidence of GIH using appropriate methods, including Chi-square tests for categorical variables and Kaplan-Meier survival analysis for cumulative hyperglycemia-free days. All analyses will be conducted with a significance level set at p < 0.05, and SPSS v20 will be used for statistical processing.

The findings from this study could provide critical insights into the potential role of dapagliflozin in preventing GIH in high-risk hospitalized patients, improving patient outcomes, and offering a new therapeutic strategy in managing hyperglycemia associated with glucocorticoid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old admitted to the emergency department with a need for hospitalization, under the care of the Internal Medicine and Hemato-Oncology departments, from May to November 2024.
* Patients with a clinical indication for high-dose glucocorticoid use (prednisone bioequivalence >30mg/day).

Exclusion Criteria:

* Current treatment with SGLT2 inhibitors, sulfonylureas, or insulin infusion pumps.
* Contraindications for SGLT2 inhibitors: chronic kidney disease (KDIGO stage IV), acute kidney injury or disease, type 1 diabetes, suspected severe acute infection, requirement for surgery, severe urinary tract infection.
* Previous use of high-dose glucocorticoids within the last 30 days. Indication for aggressive fluid resuscitation, use of vasopressors, use of mineralocorticoids, requirement for invasive mechanical ventilation, or classified as critically ill.
* Uncontrolled hyperglycemia (>140mg/dL despite proper treatment) or suspected euglycemic diabetic ketoacidosis.
* Use of glucocorticoids in the past 28 days with doses higher than medium doses (prednisone equivalence >10mg and <30mg/day).
* Inability to take dapagliflozin orally.
* Pregnancy, postpartum, or lactation.
* Patients with incomplete follow-up or inadequate adherence to the intervention protocol, or those who experience adverse effects related to dapagliflozin use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of glucocorticoid-induced hyperglycemia | until hospital discharge, an average of 10 days
  HIG (Severe Intermittent Hyperglycemia): Defined as the persistence of ≥2 events of capillary or central glucose ≥140mg/dL (7.8 mmol/L) within 24 hours.
hyperglycemia crisis | until hospital discharge, an avarage of 10 days
  Hyperglycemic Crisis (HC): Defined as the persistence of ≥2 events of capillary or central glucose ≥180mg/dL (>10 mmol/L) within 24 hours.

SECONDARY OUTCOMES:
incidence of insulin therapy. | until hospital discharge, an average of 10 days
  To determine the incidence (%) of insulin therapy use in both study arms.
Report adverse events. | until hospital dischargte, an average of 10 days
  Report adverse events associated (%) with dapagliflozin use in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Lauro F Amador Medina, Dr, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unidad Medica de Alta Especialidad Hospital de Especialidades No. 1 CMN Bajio, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
It depends on whether participants choose to share their data with other researchers outside the protocol and informed consent for this study.